CLINICAL TRIAL: NCT06674174
Title: Effects of Lower Limb Resistance Versus Endurance Training on Pulmonary Function in Smokers With Shortness of Breath
Brief Title: Effect of Lower Limb Resistance Versus Endurance Training in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Masroor Alam
Record Dates: First submitted 2024-08-13; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Endurance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lower limb strength training (Experimental): Experimental group will receive lower limb strength training
  Interventions: Other: lower limb strength training
- endurance training (Other): control group will receive endurance training.
  Interventions: Other: endurance training

INTERVENTIONS:
Other: lower limb strength training — Experimental group will receive lower limb strength training treatment for three days a week and each session will last for an hour for 3 consecutivemonths. Measurement will be recorder pre-treatment and post treatment of both groupsat baseline,3rd, and 6th week.
  Arms: lower limb strength training
Other: endurance training — Control group will receive endurance training, treatment for three days a week and each session will last for an hour for 3 consecutivemonths. Measurement will be recorder pre-treatment and post treatment of both groupsat baseline,3rd, and 6th week.
  Arms: endurance training

SUMMARY:
Patients was selected based on inclusion and exclusion criteria. Experimental group was treated with Resistance training while control group received endurance training. Data was collected by spirometry and International Physical activity questionnaire readings was recorded in every session for baseline, 3rd week and 6thweeks.

DETAILED DESCRIPTION:
Experimental group will receive lower limb strength training and control group will receive endurance training. Both groups will receive treatment for three days a week and each session will be given according to FITT formula. Measurement will be recorder pre-treatment and post treatment of both groups at baseline, third , and 6 th week.

ELIGIBILITY:
Inclusion Criteria:

* Young cigarette smokers (10 cigarette/day for at least 10 years)
* Male
* Age 25-45 years
* Sedentary lifestyle
* Body mass: less than 80kg
* BMI:22-30

Exclusion Criteria:

* Heart or pulmonary disease
* MSK disorder
* incapable of realizing the protocol of exercises,
* Recent surgery
* Recent Trauma.
* Any infective respiratory illness.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Spirometry | 6 weeks
  Spirometry is one of the Pulmonary Function Test; they are useful investigations in the management of patients with respiratory disease or respiratory weakness secondary to neurological impairment. They aid diagnosis, help monitor response to treatment and can guide decisions regarding further treatment and intervention. Spirometry can measure all the lung volumes except residual volume.
International Physical Activity Questionnaire | 6 weeks
  The International Physical Activity Questionnaire is a 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old. The International Physical Activity Questionnaire can be used clinically and in population research that compares physical activity levels between populations internationally.To calculate MET minutes a week multiply the MET value given (remember walking = 3.3, moderate activity = 4, vigorous activity = 8) by the minutes the activity was carried out and again by the number of days that that activity was undertaken. For example if someone reports walking for 30 minutes 5 days a week then the total MET minutes for that activity are 3.3 X 30 X 5=495 Met minutes a week.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Razzaq, MsCPPT, Principal Investigator — Riphah International University
Locations (1):
- Samina International Hospital, Dera Ismāīl Khān, Pakistan

IPD SHARING:
Plan to Share IPD: No